CLINICAL TRIAL: NCT02331342
Title: Comparison of NICOM and Innocor for Non-Invasive Determination of Cardiac Output
Status: Completed | Type: Observational
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Joachim Saur, senior physician, Universitätsmedizin Mannheim
Other Study IDs: NICOM IGR
Record Dates: First submitted 2015-01-02; First posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Cardiac Disease
Keywords: Agreement of NICOM and Innocor
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: NICOM cardiac output measurement
Device: Innocor cardiac output measurement

SUMMARY:
Cardiac output (CO) is an important parameter in the diagnosis and therapy of cardiac diseases. The aim of the study at hand was to evaluate NICOM (bioreactance) as a new method for determinion of CO and to compare it to Innocor (inert gas rebreathing), which previously showed promising results.

ELIGIBILITY:
Inclusion Criteria:

* hemodynamic stability
* respiratory stability

Exclusion Criteria:

* patient unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: inpatients and outpatients
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Accuracy of NICOM and Innocor | at time of inclusion
Precision of NICOM and Innocor | at time of inclusion